CLINICAL TRIAL: NCT01001377
Title: A Randomized, Multicenter, Open-label, Phase 3 Study to Compare the Efficacy and Safety of Panitumumab and Cetuximab in Subjects With Previously Treated, Wild-type KRAS, Metastatic Colorectal Cancer
Brief Title: ASPECCT: A Study of Panitumumab Efficacy and Safety Compared to Cetuximab in Patients With KRAS Wild-Type Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080763; ASPECCT; 2009-010715-32 (EudraCT Number)
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Panitumumab; Vectibix; Colon Cancer; Colorectal Cancer; Rectal Cancer; Cetuximab; Erbitux; Metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Neoplasm Metastasis | interventions — Cetuximab; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab (Active Comparator): Cetuximab 400 mg/m^2 as an initial dose, followed by 250 mg/m^2 intravenously (IV) every 7 days.
  Participants were treated until disease progression, intolerability, withdrawal of consent, or death.
  Interventions: Drug: Cetuximab
- Panitumumab (Experimental): Panitumumab 6 mg/kg IV every 14 days. Participants were treated until disease progression, intolerability, withdrawal of consent, or death.
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Cetuximab — Administered by intravenous infusion
  Other Names: Erbitux
  Arms: Cetuximab
Drug: Panitumumab — Administered by intravenous infusion
  Other Names: Vectibix
  Arms: Panitumumab

SUMMARY:
The primary objective of this study is to compare the effect of panitumumab versus cetuximab on overall survival (OS) for chemorefractory metastatic colorectal cancer (mCRC) among patients with wild-type Kirsten rat Sarcoma-2 virus (KRAS) tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the colon or rectum, metastatic disease
* Wild-type KRAS tumor status
* Eastern Cooperative Oncology Group (ECOG) score of 0, 1 or 2
* Must have failed a prior regimen containing irinotecan for metastatic disease and a prior regimen containing oxaliplatin for metastatic disease
* Must have previously received a thymidylate synthase inhibitor (eg, fluorouracil, capecitabine, raltitrexed, or fluorouracil-uracil) at any point for treatment of colorectal cancer (CRC)
* Adequate hematologic, renal, hepatic and metabolic function

Exclusion Criteria:

* Symptomatic brain metastases requiring treatment
* Prior anti-epidermal growth factor receptor (EGFr) antibody therapy (eg, panitumumab or cetuximab) or treatment with small molecule EGFr inhibitors (eg, gefitinib, erlotinib, lapatinib)
* Antitumor therapy (eg, chemotherapy, hormonal therapy, immunotherapy, antibody therapy, radiotherapy), or investigational agent or therapy ≤ 30 days before randomization.
* Clinically significant cardiovascular disease
* Active infection requiring systemic treatment or any uncontrolled infection ≤14 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2010-02-02 (Actual); Primary Completion 2013-02-05 (Actual); Study Completion 2017-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (127):
- United States (5):
  - Research Site, Stockton, California
  - Research Site, Boynton Beach, Florida
  - Research Site, Wichita, Kansas
  - Research Site, Temple, Texas
  - Research Site, Ogden, Utah
- Australia (11):
  - Research Site, Liverpool, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Wahroonga, New South Wales
  - Research Site, Wollongong, New South Wales
  - Research Site, Woodville South, South Australia
  - Research Site, Ballarat, Victoria
  - Research Site, Box Hill, Victoria
  - Research Site, Epping, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Heidelberg, Victoria
  - Research Site, Parkville, Victoria
- Research Site, Edegem, Belgium
- Research Site, Sofia, Bulgaria
- Canada (2):
  - Research Site, Edmonton, Alberta
  - Research Site, Halifax, Nova Scotia
- China (13):
  - Research Site, Guangzhou, Guangdong
  - Research Site, Harbin, Heilongjiang
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Xi'an, Shaanxi
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Chongqing, Sichuan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Beijing
  - Research Site, Shanghai
  - Research Site, Tianjin
- Czechia (6):
  - Research Site, Hořovice
  - Research Site, Nová Ves pod Pleší
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Příbram
  - Research Site, Znojmo
- France (5):
  - Research Site, Besançon
  - Research Site, Montbéliard
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Herblain
  - Research Site, Villejuif
- Hong Kong (2):
  - Research Site, Kowloon
  - Research Site, New Territories
- India (9):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Kochi, Kerala
  - Research Site, Ahilyanagar, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Nashik, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Kolkata, West Bengal
- Israel (5):
  - Research Site, Beersheba
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Ramat Gan
  - Research Site, Rehovot
- Italy (10):
  - Research Site, Ancona
  - Research Site, Cesena
  - Research Site, Cremona
  - Research Site, Faenza RA
  - Research Site, Genova
  - Research Site, Lugo
  - Research Site, Meldola FC
  - Research Site, Ravenna
  - Research Site, Rimini
  - Research Site, Torino
- Latvia (2):
  - Research Site, Daugavpils
  - Research Site, Riga
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Malaysia (3):
  - Research Site, Kota Bharu, Kelantan
  - Research Site, Kuala Lumpur, Kuala Lumpur
  - Research Site, Kota Kinabalu, Sabah
- Research Site, Rotterdam, Netherlands
- Research Site, Lima, Peru
- Philippines (3):
  - Research Site, Cebu City
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (6):
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Jelenia Góra
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Sibiu
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Serbia (2):
  - Research Site, Kamenitz
  - Research Site, Niš
- Research Site, Singapore, Singapore
- Slovakia (3):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Nitra
- South Africa (5):
  - Research Site, Groenkloof, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Kraaifontein, Western Cape
  - Research Site, Johannesburg
  - Research Site, Port Elizabeth
- South Korea (2):
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Seoul
- Sweden (6):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Uppsala
  - Research Site, Vaxjo
  - Research Site, Västerås
- Taiwan (5):
  - Research Site, Putzu City, Chiayi
  - Research Site, Keelung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (11):
  - Research Site, Belfast
  - Research Site, Bristol
  - Research Site, Cardiff
  - Research Site, Guildford
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Maidstone
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Sutton
  - Research Site, Wolverhampton

REFERENCES:
- [Background] Price T, Kim TW, Li J, Cascinu S, Ruff P, Suresh AS, Thomas A, Tjulandin S, Guan X, Peeters M. Final results and outcomes by prior bevacizumab exposure, skin toxicity, and hypomagnesaemia from ASPECCT: randomized phase 3 non-inferiority study of panitumumab versus cetuximab in chemorefractory wild-type KRAS exon 2 metastatic colorectal cancer. Eur J Cancer. 2016 Nov;68:51-59. doi: 10.1016/j.ejca.2016.08.010. Epub 2016 Oct 5. PMID 27716478
- [Background] Price TJ, Peeters M, Kim TW, Li J, Cascinu S, Ruff P, Suresh AS, Thomas A, Tjulandin S, Zhang K, Murugappan S, Sidhu R. Panitumumab versus cetuximab in patients with chemotherapy-refractory wild-type KRAS exon 2 metastatic colorectal cancer (ASPECCT): a randomised, multicentre, open-label, non-inferiority phase 3 study. Lancet Oncol. 2014 May;15(6):569-79. doi: 10.1016/S1470-2045(14)70118-4. Epub 2014 Apr 14. PMID 24739896
- [Background] Kim TW, Peeters M, Thomas A, Gibbs P, Hool K, Zhang J, Ang AL, Bach BA, Price T. Impact of Emergent Circulating Tumor DNA RAS Mutation in Panitumumab-Treated Chemoresistant Metastatic Colorectal Cancer. Clin Cancer Res. 2018 Nov 15;24(22):5602-5609. doi: 10.1158/1078-0432.CCR-17-3377. Epub 2018 Jun 13. PMID 29898991
- [Background] Peeters M, Price T, Boedigheimer M, Kim TW, Ruff P, Gibbs P, Thomas A, Demonty G, Hool K, Ang A. Evaluation of Emergent Mutations in Circulating Cell-Free DNA and Clinical Outcomes in Patients with Metastatic Colorectal Cancer Treated with Panitumumab in the ASPECCT Study. Clin Cancer Res. 2019 Feb 15;25(4):1216-1225. doi: 10.1158/1078-0432.CCR-18-2072. Epub 2018 Nov 28. PMID 30487126
- [Background] Price T, Ang A, Boedigheimer M, Kim TW, Li J, Cascinu S, Ruff P, Satya Suresh A, Thomas A, Tjulandin S, Peeters M. Frequency of S492R mutations in the epidermal growth factor receptor: analysis of plasma DNA from patients with metastatic colorectal cancer treated with panitumumab or cetuximab monotherapy. Cancer Biol Ther. 2020 Oct 2;21(10):891-898. doi: 10.1080/15384047.2020.1798695. Epub 2020 Oct 7. PMID 33026965
- [Derived] Taniguchi H, Yamanaka T, Sakai D, Muro K, Yamazaki K, Nakata S, Kimura H, Ruff P, Kim TW, Peeters M, Price T. Efficacy of Panitumumab and Cetuximab in Patients with Colorectal Cancer Previously Treated with Bevacizumab; a Combined Analysis of Individual Patient Data from ASPECCT and WJOG6510G. Cancers (Basel). 2020 Jun 28;12(7):1715. doi: 10.3390/cancers12071715. PMID 32605298
- [Derived] Graham CN, Maglinte GA, Schwartzberg LS, Price TJ, Knox HN, Hechmati G, Hjelmgren J, Barber B, Fakih MG. Economic Analysis of Panitumumab Compared With Cetuximab in Patients With Wild-type KRAS Metastatic Colorectal Cancer That Progressed After Standard Chemotherapy. Clin Ther. 2016 Jun;38(6):1376-1391. doi: 10.1016/j.clinthera.2016.03.023. Epub 2016 Apr 13. PMID 27085587
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on 2nd February 2010 and last patient enrolled 19 July 2012.
  Results are reported as of the data cut-off date of 5 February 2013.
Groups:
- Cetuximab: Cetuximab 400 mg/m^2 as an initial dose, followed by 250 mg/m^2 intravenously (IV) every 7 days.
- Panitumumab: Panitumumab 6 mg/kg IV every 14 days.
Period: Overall Study
Arm/Group | Cetuximab | Panitumumab
Started | 504 | 506
Received Treatment | 500 | 499
Completed | 78 (Indicates participants continuing in study) | 85 (Indicates participants continuing in study)
Not Completed | 426 | 421
Not completed — Ineligibility determined | 2 | 0
Not completed — Withdrawal by Subject | 19 | 20
Not completed — Lost to Follow-up | 14 | 17
Not completed — Death | 391 | 384

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab | Panitumumab | Total
Number analyzed (Participants) | 504 | 506 | 1010
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (11.2) | 59.6 (10.9) | 59.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 187 | 370
  Male | 321 | 319 | 640
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 230 | 225 | 455
  Black or African American | 4 | 2 | 6
  Hispanic or Latino | 7 | 6 | 13
  Japanese | 0 | 1 | 1
  Other | 3 | 2 | 5
  White or Caucasian | 260 | 270 | 530
Geographic region [Number; unit: participants] — Stratification factor. Rest of world includes South America, Asia and South Africa
  participants
    North America, Western Europe and Australia | 158 | 158 | 316
    Rest of World | 346 | 348 | 694
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — 0 = Fully active, able to carry on all pre-disease performance without restriction.
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, ie, light housework or office work.
  2. = Ambulatory and capable of all self-care but unable to carry out any work. activities. Up and about > 50% of waking hours.
  3. = Capable of only limited self-care, confined to a bed or chair > 50% of waking hours.
  4. = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. = Dead.
  participants
    Grade 0 | 165 | 155 | 320
    Grade 1 | 299 | 309 | 608
    Grade 2 | 40 | 42 | 82

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is the time from the date of randomization until the date of death. Participants who had not died by the analysis data cut-off date were censored at their last contact date.
Time Frame: From randomization until the data cut-off date of 5 February 2013. Maximum time on study was 155 weeks.
Population: Primary Analysis Set: All participants who were randomized and who received at least 1 dose of panitumumab or cetuximab; analyzed according to randomized treatment arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 500 | 499
months | 10.0 [9.3 to 11.0] | 10.4 [9.4 to 11.6]
Statistical Analysis 1: Comparison: Cetuximab vs Panitumumab; Cox proportional hazards model stratified by geographic region (North America, western Europe and Australia vs rest of world) and ECOG performance status (0 or 1 vs 2); Test type: Superiority or Other; Stratified Cox proportional hazard ratio = 0.966, 95% CI 2-sided [0.839 to 1.113] — Hazard ratio is presented as panitumumab : cetuximab. A value < 1.0 indicates a lower average event rate and longer time to event for panitumumab relative to cetuximab
Statistical Analysis 2: Comparison: Cetuximab vs Panitumumab; A synthesis approach with an asymptotic standard normal test statistic based on the logarithm of the hazard ratio was used to test the hypothesis that panitumumab is non-inferior to cetuximab for overall survival (ie, that panitumumab retains at least 50% of the overall survival benefit of cetuximab relative to best supportive care); Test type: Non-Inferiority or Equivalence — The overall survival non-inferiority hypothesis based on an asymptotic normal score was tested at a 1-sided 2.5% significance level. A value < -1.96 indicates non-inferiority at a significance level of 1-sided 0.025; p = 0.0007, Asymptotic standard normal test — A synthesis approach with an asymptotic standard normal test statistic; Normal score = -3.19

2. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is the time from the date of randomization to the date of disease progression per the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 or death. Participants alive and not meeting criteria for progression by the analysis data cut-off date were censored at their last evaluable disease assessment date.
  Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study based on all target lesions recorded since the treatment started (the sum must also demonstrate an absolute increase of at least 5 mm), or unequivocal progression of existing non-target lesions, or any new lesions.
Time Frame: From randomization until the data cut-off date of 5 February 2013. Maximum time on study was 155 weeks.
Population: Primary analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 500 | 499
months | 4.4 [3.2 to 4.8] | 4.1 [3.2 to 4.8]

3. Secondary Outcome: Objective Response
Description: Objective response is either a complete response (CR) or partial response (PR) per RECIST version 1.1. All participants that did not meet the criteria for an objective response by the analysis cut-off date were considered non-responders. CR: Disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm, and disappearance of all non-target lesions, and no new lesions. PR: Disappearance of all target lesions, persistence of one or more non-target lesions not qualifying for either CR or progressive disease, or, at least a 30% decrease in the sum of diameters of target lesions with no unequivocal progression of existing non-target lesions and no new lesions.
Time Frame: From randomization until the data cut-off date of 5 February 2013. Maximum time on study was 155 weeks.
Population: Tumor Response Analysis Set: Participants in the primary analysis set with at least 1 Baseline unidimensionally measurable lesion per RECIST version 1.1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 485 | 486
percentage of participants | 19.79 [16.34 to 23.62] | 22.02 [18.41 to 25.97]
Statistical Analysis 1: Comparison: Cetuximab vs Panitumumab; Test type: Superiority or Other; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.83 to 1.58] — Common treatment odds ratio stratified by geographic region (North America, western Europe and Australia vs rest of world) and ECOG performance status (0 or 1 vs 2)

4. Secondary Outcome: Duration of Response
Description: Duration of response (DOR), calculated only for those participants with an objective response, is the time from first objective response to disease progression per the RECIST v1.1 or death. Participants not meeting criteria for progression or who died by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Time Frame: From randomization until the data cut-off date of 5 February 2013. Maximum time on study was 155 weeks.
Population: Participants with an objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 96 | 107
months | 5.4 [3.8 to 5.5] | 3.8 [3.7 to 4.8]

5. Secondary Outcome: Time to Response
Description: Time to response (TTR), calculated for those participants with an objective response, is defined as the time from the randomization date to the date of first objective response.
Time Frame: From randomization until the data cut-off date of 5 February 2013. Maximum time on study was 155 weeks.
Population: Participants with an objective response
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 96 | 107
months | 2.6 [1.2 to 3.1] | 1.5 [1.2 to 3.0]

6. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure (TTF) is the time from randomization date to date that the decision was made to end the treatment period for any reason; participants who remained in the treatment period at the time of analysis were censored at the date of the last on-study assessment.
Time Frame: From randomization until the data cut-off date of 5 February 2013. Maximum time on study was 155 weeks.
Population: Primary analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 500 | 499
months | 3.3 [3.2 to 3.9] | 3.4 [3.2 to 4.6]

7. Secondary Outcome: Change From Baseline in EuroQOL 5 Dimension (EQ-5D) Health State Index Score
Description: The EQ-5D is a standardized instrument for use as a generic measure of health outcome. The health state index measures the following 5 health dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension contains 3 levels of response to reflect degree of problems participants have experienced: no problem (1), some problem (2) and extreme problems (3). The health states for each respondent are converted into a single index number using a specified set of weights. Resulting scores can range from 1.0 and -0.594. A higher score indicates a more preferred health status with 1.0 representing perfect health and 0 representing death. Negative scores are possible and represent health states regarded as less preferable than death (0). Repeated measures mixed model includes treatment, geographic region, ECOG score, assessment week, and treatment by assessment week interaction as fixed effects, and participants a random effect.
Time Frame: From Study Day 1 through the last day of treatment or disease progression, up to Week 85.
Population: Patient reported outcomes (PRO) analysis set: all participants in the primary analysis set who have a Baseline and at least one follow-up PRO assessment prior to clinical or objective disease progression per RECIST version 1.1. Participants with available data are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 150 | 143
scores on a scale | -0.0341 [-0.0806 to 0.0123] | -0.0216 [-0.0691 to 0.0260]
Statistical Analysis 1: Comparison: Cetuximab vs Panitumumab; Repeated measures mixed model includes treatment, geographic region, ECOG score, assessment week, and treatment by assessment week interaction as fixed effects, and subjects a random effect. An unstructured covariance matrix is used in the mixed model; Test type: Superiority or Other; LS Mean Difference = 0.0126, 95% CI 2-sided [-0.0353 to 0.0605] — A positive difference between the treatment groups favors the panitumumab group

8. Secondary Outcome: Change From Baseline in EuroQOL 5 Dimension (EQ-5D) Visual Analog Scale (VAS)
Description: The EQ-5D is a standardized instrument for use as a generic measure of health outcome. The VAS asks respondents to rate their present health status on a 0 - 100 scale, with 0 labeled as "Worst imaginable health state" and 100 labeled as "Best imaginable health state." The VAS score is determined by observing the point at which the participant's hand drawn line intersects the scale.
Time Frame: From Study Day 1 through the last day of treatment or disease progression, up to Week 85.
Population: Patient reported outcomes (PRO) analysis set participants with available data
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 149 | 142
scores on a scale | 3.9782 [0.8842 to 7.0722] | 2.3037 [-0.8532 to 5.4605]
Statistical Analysis 1: Comparison: Cetuximab vs Panitumumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -1.6745, 95% CI 2-sided [-4.9331 to 1.5841] — A positive difference between the treatment groups favors the panitumumab group

9. Secondary Outcome: Change From Baseline in National Comprehensive Cancer Network Functional Assessment of Cancer Therapy Colorectal Symptom Index (NCCN FCSI ) Symptoms Score
Description: The FCSI consists of 9 questions comprising the most important symptoms associated with colorectal cancer, including energy, pain, weight, diarrhea, nausea, swelling or cramps in the stomach area, appetite, ability to enjoy life, and overall quality of life. The 9 questions are combined in three algorithms to provide information for 3 domains: colorectal cancer symptoms, physical well-being, and functional well-being. Each of the 9 items are scored from "0" to "4" representing "Not at All" through to "Very Much True". The raw score for all items is transformed to a 0-100 scale, and the average for each of the 3 subscales is calculated; high scores illustrate an improved state (e.g. able to enjoy life more).
Time Frame: From Study Day 1 through the last day of treatment or disease progression, up to Week 85.
Population: Patient reported outcomes (PRO) analysis set participants with available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 151 | 142
scores on a scale | 2.0101 [-1.1477 to 5.1679] | 3.0473 [-0.1782 to 6.2728]
Statistical Analysis 1: Comparison: Cetuximab vs Panitumumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 1.0372, 95% CI 2-sided [-2.3267 to 4.4010] — A positive difference between the treatment groups favors the panitumumab group

10. Secondary Outcome: Change From Baseline in NCCN FCSI Physical Well-being Scale Score
Description: as for outcome 9
Time Frame: From Study Day 1 through the last day of treatment or disease progression, up to Week 85.
Population: Patient reported outcomes (PRO) analysis set participants with available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 150 | 142
scores on a scale | 1.8778 [-1.5524 to 5.3080] | 2.4614 [-1.0442 to 5.9670]
Statistical Analysis 1: Comparison: Cetuximab vs Panitumumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 0.5836, 95% CI 2-sided [-3.0269 to 4.1941] — A positive difference between the treatment groups favors the panitumumab group

11. Secondary Outcome: Change From Baseline in NCCN FCSI Functional Well-being Scale Score
Description: as for outcome 9
Time Frame: From Study Day 1 through the last day of treatment or disease progression, up to Week 85.
Population: Patient reported outcomes (PRO) analysis set participants with available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 152 | 143
scores on a scale | 1.3567 [-4.1564 to 6.8697] | 1.1569 [-4.4887 to 6.8025]
Statistical Analysis 1: Comparison: Cetuximab vs Panitumumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -0.1998, 95% CI 2-sided [-6.0093 to 5.6098] — A positive difference between the treatment groups favors the panitumumab group

12. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Serious adverse events include any event that is fatal, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or other significant medical hazard. Treatment-related AEs are those the investigator considered as a reasonable possibility to have been caused by study drug.
Time Frame: From the day of the first dose of study therapy through 30 days since the last dose. Maximum time on study treatment was 130 weeks.
Population: Safety Analysis Set (randomized participants who received at least 1 dose of study medication). Five participants who received the incorrect study medication (4 assigned to panitumumab but received cetuximab and 1 assigned to cetuximab but received panitumumab) were included in different treatment arms for safety analyses.
Measure: Number; unit: participants
Arm/Group | Cetuximab | Panitumumab
Number analyzed (Participants) | 503 | 496
participants
  Any adverse event (AE) | 494 | 485
  Serious adverse events | 169 | 151
  Leading to discontinuation of study drug | 61 | 69
  Any treatment-related adverse event (TRAE) | 459 | 437
  Treatment-related serious adverse event | 22 | 25
  TRAE leading to discontinuation of study drug | 15 | 14

ADVERSE EVENTS:
Time Frame: Median time was 117 days for panitumumab arm and 123 days for cetuximab arm.
Description: Five participants who received the incorrect study medication (4 assigned to panitumumab but received cetuximab and 1 assigned to cetuximab but received panitumumab) were included in different treatment arms for safety analyses.
  The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Cetuximab | Panitumumab
Serious Adverse Events (participants affected / at risk) | 169/503 | 151/496
Other Adverse Events (participants affected / at risk) | 474/503 | 459/496
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=503) | Panitumumab (N=496)
Anaemia (Blood and lymphatic system disorders) | 3 | 6
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 10
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Ascites (Gastrointestinal disorders) | 5 | 5
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 8 | 6
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 5 | 5
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 8 | 12
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 2
Obturator hernia (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 4
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 5 | 12
Asthenia (General disorders) | 4 | 6
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Device occlusion (General disorders) | 0 | 2
Fatigue (General disorders) | 4 | 4
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 2 | 1
Hyperpyrexia (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 1
Pain (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 1
Pyrexia (General disorders) | 8 | 3
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 2 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 2
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 1
Jaundice (Hepatobiliary disorders) | 0 | 3
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 0
Jaundice extrahepatic obstructive (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 3 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 2
Cystitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 2
Device related sepsis (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 2
Lobar pneumonia (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 2 | 0
Nail infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 1
Pyonephrosis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 5
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary bladder abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 7 | 9
Urosepsis (Infections and infestations) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 2
Blood creatine increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Blood uric acid increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 2
Red blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 7
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 7
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 2 | 0
Bladder dilatation (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 4
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 2
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 2
Ureteric stenosis (Renal and urinary disorders) | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Central venous catheterisation (Surgical and medical procedures) | 0 | 1
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 0 | 1
Artery dissection (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=503) | Panitumumab (N=496)
Anaemia (Blood and lymphatic system disorders) | 30 | 29
Abdominal pain (Gastrointestinal disorders) | 74 | 52
Constipation (Gastrointestinal disorders) | 70 | 39
Diarrhoea (Gastrointestinal disorders) | 87 | 88
Dyspepsia (Gastrointestinal disorders) | 26 | 19
Nausea (Gastrointestinal disorders) | 56 | 66
Stomatitis (Gastrointestinal disorders) | 34 | 26
Vomiting (Gastrointestinal disorders) | 49 | 49
Asthenia (General disorders) | 44 | 30
Fatigue (General disorders) | 85 | 72
Oedema peripheral (General disorders) | 38 | 22
Pyrexia (General disorders) | 50 | 28
Paronychia (Infections and infestations) | 75 | 58
Upper respiratory tract infection (Infections and infestations) | 28 | 14
Weight decreased (Investigations) | 21 | 26
Decreased appetite (Metabolism and nutrition disorders) | 77 | 69
Hypocalcaemia (Metabolism and nutrition disorders) | 16 | 26
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 41
Hypomagnesaemia (Metabolism and nutrition disorders) | 89 | 134
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 34
Headache (Nervous system disorders) | 36 | 17
Insomnia (Psychiatric disorders) | 46 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 40
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 19
Acne (Skin and subcutaneous tissue disorders) | 69 | 52
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 136 | 138
Dry skin (Skin and subcutaneous tissue disorders) | 79 | 83
Nail disorder (Skin and subcutaneous tissue disorders) | 31 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 88 | 83
Rash (Skin and subcutaneous tissue disorders) | 257 | 249
Skin fissures (Skin and subcutaneous tissue disorders) | 43 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.